CLINICAL TRIAL: NCT06451133
Title: Hemodynamic Management Following Acute Traumatic Spinal Cord Injury: A Randomized, Controlled Trial
Brief Title: Hemodynamic Management Following Acute Traumatic Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Trauma Research and Combat Casualty Care Collaborative (TRC4) (Unknown)
Responsible Party: Principal Investigator, David E. Meyer, MD, MS, FACS, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-24-0405
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mean arterial blood pressure (MAP) goal of ≥65 mmHg (Experimental)
  Interventions: Other: Mean arterial blood pressure (MAP) goal of ≥65 mmHg
- Mean arterial blood pressure (MAP) goal of 85-90 mmHg (Experimental)
  Interventions: Other: Mean arterial blood pressure (MAP) goal of 85-90 mmHg
- Spinal cord perfusion pressure (SCPP) goal of ≥65 mmHg (Experimental)
  Interventions: Other: Spinal cord perfusion pressure (SCPP) goal of ≥65 mmHg

INTERVENTIONS:
Other: Mean arterial blood pressure (MAP) goal of ≥65 mmHg — The treatment team will maintain MAP ≥65 mmHg for the first five days following injury.
  Arms: Mean arterial blood pressure (MAP) goal of ≥65 mmHg
Other: Mean arterial blood pressure (MAP) goal of 85-90 mmHg — The treatment team will maintain MAP 85-90 mmHg for the first five days following injury.
  Arms: Mean arterial blood pressure (MAP) goal of 85-90 mmHg
Other: Spinal cord perfusion pressure (SCPP) goal of ≥65 mmHg — The treatment team will maintain SCPP ≥65 mmHg for the first five days following injury.
  Arms: Spinal cord perfusion pressure (SCPP) goal of ≥65 mmHg

SUMMARY:
The purpose of this study is to assess the effect of various hemodynamic management strategies on functional neurologic outcomes and non-neurologic adverse events in the first 5 days following acute spinal cord injury (SCI). The hemodynamic management strategies assessed include targeting a mean arterial blood pressure (MAP) goal of 85-90 mmHg, targeting a spinal cord perfusion pressure (SCPP) goal of ≥65 mmHg, or targeting normal hemodynamics, which is a MAP goal of ≥65 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic spinal cord injury

Exclusion Criteria:

* Patients with an injury from a trauma that penetrates the spinal cord (i.e., gunshot or knife wound resulting in cord transection)
* Preexisting neurologic or spinal cord injury
* Severe traumatic brain injury as measured by a best resuscitated Glasgow Coma Scale (GCS) score of <8 at 24 hours following injury
* Presence of traumatic injuries that preclude spine surgery within 24 hours of presentation
* Concomitant injury/illness requiring targeted blood pressure management (e.g., injury to the aorta, aortic dissection, hemorrhagic stroke)
* Preexisting history of neuromotor disorders (i.e., cerebral palsy, Parkinson disease, etc.)
* Not expected to survive >24h
* Cord transection identified by radiologist and agreed upon by the spine surgery team
* Injury below spinal cord level L1
* Prisoners
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The severity of a spinal cord injury (SCI) as assessed by the American Spinal Injury Association (ASIA) International Standards for Neurological Classification of Spinal Cord Injury (ISNCSC) motor score | 6 weeks following injury
  Upper and lower extremities will be assessed, and motor strength at each spinal cord level will be scored from 0 to 5 (0 indicates total paralysis and 5 indicates active movement against full resistance), with a maximum score of 25 for each extremity, totaling 100 for all four extremities. Total score ranges from 0 to 100, with a higher score indicating a better outcome.
Performance in activities of daily living and mobility as assessed by the Spinal Cord Independence Measure (SCIM) III score | 6 weeks following injury
  There are 3 subscales on the SCIM III: self-care (4 items, score ranging from 0-20), respiration and sphincter management (4 items, score ranging from 0-40), and mobility (9 items, score ranging from 0-40). Total score ranges from 0 to 100, with a higher score indicating a better outcome.

SECONDARY OUTCOMES:
Change in motor function as assessed by the American Spinal Injury Association (ASIA) International Standards for Neurological Classification of Spinal Cord Injury (ISNCSC) motor score | 6 months following injury, 12 months following injury
  Upper and lower extremities will be assessed, and motor strength at each spinal cord level will be scored from 0 to 5 (0 indicates total paralysis and 5 indicates active movement against full resistance), with a maximum score of 25 for each extremity, totaling 100 for all four extremities. Total score ranges from 0 to 100, with a higher score indicating a better outcome.
Change in sensory function as assessed by the American Spinal Injury Association (ASIA) International Standards for Neurological Classification of Spinal Cord Injury (ISNCSC) sensory score | 6 months following injury, 12 months following injury
  For each side of the body, 28 key sensory points will be assessed by light touch, and each area will be scored from 0 to 2 (0 indicates sensing is absent, 1 indicates sensing is altered, and 2 indicates that sensing is normal). Additionally, for each side of the body 28 key sensory points will be also be assessed by pin prick, and each area will be scored from 0 to 2 (0 indicates sensing is absent, 1 indicates sensing is altered, and 2 indicates that sensing is normal). Scores for light touch and pin prick assessments for both sides of the body will be combined, and the total score ranges from 0 to 224, with a higher score indicating a better outcome.
Change in performance in activities of daily living and mobility as assessed by the Spinal Cord Independence Measure (SCIM) III score | 6 months following injury, 12 months following injury
  There are 3 subscales on the SCIM III: self-care (4 items, score ranging from 0-20), respiration and sphincter management (4 items, score ranging from 0-40), and mobility (9 items, score ranging from 0-40). Total score ranges from 0 to 100, with a higher score indicating a better outcome.
Number of ICU-free days | 30 days from baseline
  Number of ICU-free days = [30 days - ICU length of stay in days]. Patients with ICU length of stay >30 days will be assigned a value of zero ICU-free days.
Duration of time (hours) receiving goal caloric requirements by enteric nutrition | first 5 days of hospitalization
Number of participants developing a central line-associated blood stream infection | Baseline to hospital discharge or 30 days, whichever comes first
  Blood stream infection is defined as bacteremia confirmed by blood culture in the presence of a central venous catheter.
Number of participants developing a pneumothorax from central venous catheter insertion | Baseline to hospital discharge or 30 days, whichever comes first
Number of participants developing pneumonia | Baseline to hospital discharge or 30 days, whichever comes first
  Pneumonia is defined as 10,000 colony forming units (cfu)/milliliter (mL) on bronchioalveolar lavage or mini bronchioalveolar lavage, or clinical diagnosis of pneumonia with subsequent antibiotic treatment.
Number of participants developing acute kidney injury using the Risk, Injury, Failure, Loss of kidney function, and End-stage kidney disease (RIFLE) criteria | Baseline to hospital discharge or 30 days, whichever comes first
  Acute kidney injury using the RIFLE criteria is defined as a 50% increase in serum creatinine from baseline or urine output <0.5 mL/h for 6 hours.
Number of deaths | Baseline to hospital discharge or 30 days, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: David Meyer, MD, MS, FACS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No